CLINICAL TRIAL: NCT03665051
Title: Electrical Stimulation of Human Myocytes in Microgravity: An In Vitro Model to Evaluate Therapeutics to Counteract Muscle Wasting (microG)
Brief Title: Electrical Stimulation of Human Myocytes in Microgravity
Acronym: microG
Status: Active, not recruiting | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: TRIMD 1311789
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young adults: Obtain muscle biopsy specimens from young adults (ages 20-40) to develop a millifluidic chip for electrical stimulation of human primary muscle cell hydrogel cultures.
  Interventions: Procedure: Muscle Tissue Biopsy; Other: Maximal Oxygen Consumption (V02max)
- Older adults: Obtain muscle biopsy specimens from older adults (ages 60-80) to develop a millifluidic chip for electrical stimulation of human primary muscle cell hydrogel cultures.
  Interventions: Procedure: Muscle Tissue Biopsy; Other: Maximal Oxygen Consumption (V02max)

INTERVENTIONS:
Procedure: Muscle Tissue Biopsy — A biopsy of the Vastus Lateralis muscle will be performed on the left leg using the Bergstrom technique.The skin will be incised (approximately 0.75 cm) with a #11 scalpel, and the Bergstrom needle will be inserted into the Vastus Lateralis. Approximately 150 mg of muscle tissue will be obtained under suction. After the biopsy, pressure will be applied to stop bleeding and the skin will be closed with Steri strips (suture(s) if allergy to steri strips and removal 7-10 days post biopsy). A sterile dressing will be applied. Ace bandage may also be used along with applied pressure and an ice pack for any swelling and pain relief.
Other: Maximal Oxygen Consumption (V02max) — Aerobic fitness will be determined by measuring maximal O2 consumption (VO2max) during a stationary bicycle exercise test. Heart rate, blood pressure and ECG will be recorded throughout this test. Subjects will breathe through a low resistance mouthpiece and wear a nose clip. Expired gases will be measured by indirect calorimetry and heart rate monitored by a portable heart rate monitor. Following a standardized warm up, subjects will begin exercising at a moderate intensity with the workload increased every minute until the subject can no longer continue. A leveling-off (plateau) or decline in oxygen uptake should be demonstrated in order to be reasonably sure that a subject has achieved the maximum capacity for aerobic metabolism.

SUMMARY:
The purpose of this study is to evaluate the changes of muscle, in microgravity. Which will help explain the health benefits of exercise. There are tests that can be done to tell researchers more about the human body, such as a dual energy x-ray absorptiometry (DEXA) scan, which measures body composition (fat and lean body mass). The use of muscle testing and a Handgrip test can tell us about the strength and power within an individual's muscles. A VO2 max test helps us understand the aerobic fitness level of an individual and one of the most important aspects of this study are muscle cells. A muscle biopsy allows us to obtain muscle cells from the thigh, which will be sent into space by a rocket. Researchers will study these muscle cells in a low gravity environment aboard the International Space Station. Studying the muscle cells under those conditions will potentially mimic an accelerated aging process, which will help researchers better understand muscle wasting in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Participant is capable of giving informed consent and has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board and provided Health Insurance Portability and Accountability Act authorization (HIPAA) or other privacy authorization prior to any participation in study.
* Participant is 20-40 or 60-80 years of age, inclusive
* Participant BMI <30 kg/m2
* Participant states willingness to follow protocol as described, including the prescribed activity level and completing any forms needed throughout the study.

Exclusion Criteria:

* Participant reports a history of type 1 or type 2 Diabetes; or Hgb A1c > 6.5% at screening visit.
* Participant is actively pursuing weight loss and/or lifestyle changes.
* Participant has a history of pressure ulcers.
* Participant has a stated history of Deep Vein Thrombosis (DVT), recent (within last 3 months) pulmonary embolism, or has a positive D-dimer test and lower extremity ultrasound at screening, or a known hypercoagulable condition, or other clotting or bleeding disorders.
* Participant has poorly controlled hypertension or hypotension in the opinion of the study PI or medical investigator (MI).
* Participant has untreated hypothyroidism or hyperthyroidism.
* Participant has current infection (requiring prescription antimicrobial or antiviral medication, or hospitalization), or corticosteroid treatment (with the exception of inhaled or topical steroids) in the last 3 months prior to screening visit.
* Participant is currently taking prescription strength anti-inflammatory medication or has taken prescription strength anti-inflammatory medication in the 6 weeks prior to screening.
* Participant has had surgery requiring >2 days of hospitalization in the last 3 weeks prior to screening visit.
* Participant has an active malignancy or autoimmune disease.
* Participant has current significantly impaired liver function in the opinion of the study PI (mild asymptomatic fatty liver is acceptable), or hepatic enzyme tests are ≥2.5 times normal limit.
* Participant has a chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis B or C, or HIV, per self-report.
* Participant is an amputee and/or has presence of partial or full artificial limb.
* Participant has had a significant cardiovascular event (e.g. myocardial infarction, stroke) ≤ 6 months prior to screening visit; or stated history of congestive heart failure; or participant has evidence of cardiovascular disease assessed during the ECG at screening.
* Participant has a history of, or currently has uncontrolled severe diarrhea, nausea or vomiting.
* Participant has an obstruction of the gastrointestinal tract, inflammatory bowel disease, short bowel syndrome or other forms of gastrointestinal disease such as stage III or above gastroesophageal reflux disease, gastroparesis, peptic ulcer disease, celiac disease, intestinal dysmotility, diverticulitis, ischemic colitis.
* Participant has used tobacco within the last 3 months.
* Participant has a history of drug or alcohol abuse (> 3 drinks per day) within the last 5 years
* Female participant is pregnant, lactating or is within 6 weeks postpartum prior to the screening visit
* Participant has impaired renal function: estimated glomerular filtration rate (eGFR) ≤ 50 ml/min/1.73m2 determined at screening.
* Participant's triglyceride level is ≥ 250 mg/dl and LDL cholesterol is > 150 mg/dl at screening.
* Participant has a urine albumin-to-creatinine ratio (UACR) ≥300 mg/g at screening in a single urine specimen (per National Kidney Foundation guideline).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and females in the age ranges 20-40 and 60-80 years were recruited. Participants were medically screened to determine good health, weight stable (less than 3kg weight change during the previous 6 months), and without any contraindication to exercise. Approximately equal numbers of men and women were be recruited. Neither race nor ethnicity were exclusions.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-01-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Muscle biopsy parameters | About 30 minutes
  Collection of the muscle biopsy parameters (isolated satellite cells), from 9 participants in each of young and old study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Coen, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim TN, Choi KM. Sarcopenia: definition, epidemiology, and pathophysiology. J Bone Metab. 2013 May;20(1):1-10. doi: 10.11005/jbm.2013.20.1.1. Epub 2013 May 13. PMID 24524049
- [Background] Cohen S, Nathan JA, Goldberg AL. Muscle wasting in disease: molecular mechanisms and promising therapies. Nat Rev Drug Discov. 2015 Jan;14(1):58-74. doi: 10.1038/nrd4467. PMID 25549588
- [Background] Baumgartner RN, Koehler KM, Gallagher D, Romero L, Heymsfield SB, Ross RR, Garry PJ, Lindeman RD. Epidemiology of sarcopenia among the elderly in New Mexico. Am J Epidemiol. 1998 Apr 15;147(8):755-63. doi: 10.1093/oxfordjournals.aje.a009520. PMID 9554417
- [Background] Janssen I, Shepard DS, Katzmarzyk PT, Roubenoff R. The healthcare costs of sarcopenia in the United States. J Am Geriatr Soc. 2004 Jan;52(1):80-5. doi: 10.1111/j.1532-5415.2004.52014.x. PMID 14687319
- [Background] Brioche T, Lemoine-Morel S. Oxidative Stress, Sarcopenia, Antioxidant Strategies and Exercise: Molecular Aspects. Curr Pharm Des. 2016;22(18):2664-78. doi: 10.2174/1381612822666160219120531. PMID 26891808
- [Background] Fitts RH, Trappe SW, Costill DL, Gallagher PM, Creer AC, Colloton PA, Peters JR, Romatowski JG, Bain JL, Riley DA. Prolonged space flight-induced alterations in the structure and function of human skeletal muscle fibres. J Physiol. 2010 Sep 15;588(Pt 18):3567-92. doi: 10.1113/jphysiol.2010.188508. Epub 2010 Jul 26. PMID 20660569
- [Background] Trappe S, Costill D, Gallagher P, Creer A, Peters JR, Evans H, Riley DA, Fitts RH. Exercise in space: human skeletal muscle after 6 months aboard the International Space Station. J Appl Physiol (1985). 2009 Apr;106(4):1159-68. doi: 10.1152/japplphysiol.91578.2008. Epub 2009 Jan 15. PMID 19150852
- [Background] Allen DL, Bandstra ER, Harrison BC, Thorng S, Stodieck LS, Kostenuik PJ, Morony S, Lacey DL, Hammond TG, Leinwand LL, Argraves WS, Bateman TA, Barth JL. Effects of spaceflight on murine skeletal muscle gene expression. J Appl Physiol (1985). 2009 Feb;106(2):582-95. doi: 10.1152/japplphysiol.90780.2008. Epub 2008 Dec 12. PMID 19074574
- [Background] Vandenburgh H, Chromiak J, Shansky J, Del Tatto M, Lemaire J. Space travel directly induces skeletal muscle atrophy. FASEB J. 1999 Jun;13(9):1031-8. doi: 10.1096/fasebj.13.9.1031. PMID 10336885
- [Background] Higashibata A, Hashizume T, Nemoto K, Higashitani N, Etheridge T, Mori C, Harada S, Sugimoto T, Szewczyk NJ, Baba SA, Mogami Y, Fukui K, Higashitani A. Microgravity elicits reproducible alterations in cytoskeletal and metabolic gene and protein expression in space-flown Caenorhabditis elegans. NPJ Microgravity. 2016 Jan 21;2:15022. doi: 10.1038/npjmgrav.2015.22. eCollection 2016. PMID 28725720
- [Background] Aas V, Bakke SS, Feng YZ, Kase ET, Jensen J, Bajpeyi S, Thoresen GH, Rustan AC. Are cultured human myotubes far from home? Cell Tissue Res. 2013 Dec;354(3):671-82. doi: 10.1007/s00441-013-1655-1. Epub 2013 Jun 8. PMID 23749200
- [Background] Gaster M, Petersen I, Hojlund K, Poulsen P, Beck-Nielsen H. The diabetic phenotype is conserved in myotubes established from diabetic subjects: evidence for primary defects in glucose transport and glycogen synthase activity. Diabetes. 2002 Apr;51(4):921-7. doi: 10.2337/diabetes.51.4.921. PMID 11916908
- [Background] Henry RR, Ciaraldi TP, Abrams-Carter L, Mudaliar S, Park KS, Nikoulina SE. Glycogen synthase activity is reduced in cultured skeletal muscle cells of non-insulin-dependent diabetes mellitus subjects. Biochemical and molecular mechanisms. J Clin Invest. 1996 Sep 1;98(5):1231-6. doi: 10.1172/JCI118906. PMID 8787686
- [Background] Thompson DB, Pratley R, Ossowski V. Human primary myoblast cell cultures from non-diabetic insulin resistant subjects retain defects in insulin action. J Clin Invest. 1996 Nov 15;98(10):2346-50. doi: 10.1172/JCI119046. PMID 8941652
- [Background] McGregor RA, Poppitt SD, Cameron-Smith D. Role of microRNAs in the age-related changes in skeletal muscle and diet or exercise interventions to promote healthy aging in humans. Ageing Res Rev. 2014 Sep;17:25-33. doi: 10.1016/j.arr.2014.05.001. Epub 2014 May 14. PMID 24833328
- [Background] Hangelbroek RW, Fazelzadeh P, Tieland M, Boekschoten MV, Hooiveld GJ, van Duynhoven JP, Timmons JA, Verdijk LB, de Groot LC, van Loon LJ, Muller M. Expression of protocadherin gamma in skeletal muscle tissue is associated with age and muscle weakness. J Cachexia Sarcopenia Muscle. 2016 Dec;7(5):604-614. doi: 10.1002/jcsm.12099. Epub 2016 Feb 2. PMID 27239416
- [Background] Su J, Ekman C, Oskolkov N, Lahti L, Strom K, Brazma A, Groop L, Rung J, Hansson O. A novel atlas of gene expression in human skeletal muscle reveals molecular changes associated with aging. Skelet Muscle. 2015 Oct 9;5:35. doi: 10.1186/s13395-015-0059-1. eCollection 2015. PMID 26457177
- [Background] Chopard A, Lecunff M, Danger R, Lamirault G, Bihouee A, Teusan R, Jasmin BJ, Marini JF, Leger JJ. Large-scale mRNA analysis of female skeletal muscles during 60 days of bed rest with and without exercise or dietary protein supplementation as countermeasures. Physiol Genomics. 2009 Aug 7;38(3):291-302. doi: 10.1152/physiolgenomics.00036.2009. Epub 2009 May 26. PMID 19470803
- [Background] Robinson MM, Dasari S, Konopka AR, Johnson ML, Manjunatha S, Esponda RR, Carter RE, Lanza IR, Nair KS. Enhanced Protein Translation Underlies Improved Metabolic and Physical Adaptations to Different Exercise Training Modes in Young and Old Humans. Cell Metab. 2017 Mar 7;25(3):581-592. doi: 10.1016/j.cmet.2017.02.009. PMID 28273480
- [Background] Adams CM, Ebert SM, Dyle MC. Use of mRNA expression signatures to discover small molecule inhibitors of skeletal muscle atrophy. Curr Opin Clin Nutr Metab Care. 2015 May;18(3):263-8. doi: 10.1097/MCO.0000000000000159. PMID 25807353
- [Background] Dyle MC, Ebert SM, Cook DP, Kunkel SD, Fox DK, Bongers KS, Bullard SA, Dierdorff JM, Adams CM. Systems-based discovery of tomatidine as a natural small molecule inhibitor of skeletal muscle atrophy. J Biol Chem. 2014 May 23;289(21):14913-24. doi: 10.1074/jbc.M114.556241. Epub 2014 Apr 9. PMID 24719321
- [Background] Sparks LM, Moro C, Ukropcova B, Bajpeyi S, Civitarese AE, Hulver MW, Thoresen GH, Rustan AC, Smith SR. Remodeling lipid metabolism and improving insulin responsiveness in human primary myotubes. PLoS One. 2011;6(7):e21068. doi: 10.1371/journal.pone.0021068. Epub 2011 Jul 8. PMID 21760887
- See also: Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org/

DOCUMENTS (1):
  • Informed Consent Form (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT03665051/ICF_000.pdf